| Project Title: Use | r Evaluation o | of the Gui | ide To Go | als Applica | tion - a | Care C | Coordination | Tool to | Translate |
|---|---|---|---|---|---|---|---|---|---|
| | ADA Clinical | Standard | ls of Care | for Childre | en With | T2D Ir | nto Practice | | |

NCT Number: NCT03926598

Date: December 13, 2022

### **Study Protocol**

The purpose of this project was to evaluate the user interface of the Guide to Goals (GTG) application for ease-of-use. By observing and analyzing actual user experience with the current version of the app, we aimed to learn about its shortcomings. Findings from this phase will be used to make GTG application more user friendly. The GTG application was aimed at the following user groups: 1. Patients/caretakers 2. Front-desk staff 3. Nurses 4. Certified Diabetes Educators 5. Physicians. In this study, we aimed to recruit two participants from each of the five user groups for a one-hour usability testing session. However, due to limitations experienced during the COVID-19 pandemic, only 1 participant from the patient/caretaker group, 2 front desk staff, 2 nurses, 1 certified diabetes educator, and 0 physicians were enrolled, for a total of 6 participants.

The usability testing session consisted of tasks that were to be performed by the user on the GTG application, a post interview, and a post survey. The specific set of tasks that each participant was asked to perform varied between groups. The following list describes what each group was asked to do when performing the tasks on the GTG application (Note: the physician group is not described as 0 participants were enrolled from this group).

# 1. Patient and/or Family Member

- a. On the Patient Login Screen, log in using your last name and session ID provided by the research team on the Surveys Screen.
- b. Click on a pending survey when the survey opens.
- c. Respond to the survey submit the survey log out of the Guide-Goals Application

## 2. Front Desk Staff

- a. On the Provider Login Screen, log in using the username and password provided by the research team on the Patient Screen.
- b. Add a new patient on the Edit Patient Screen.
- c. Add the Diabetes Family Responsibility Questionnaire on the Edit Patient Screen.
- d. Create a survey access code to share with the patient

#### 3. Nurse

- a. On the Provider Login Screen, log in using the username and password provided by the research team on the Patients Screen.
- b. Choose patient Will Owens on the Visit Status screen.
- c. Change HbA1C value to 10% on the Visit Status screen.
- d. Change Nephropathy evaluation to Abnormal log out of Guide to Goals application.

#### 4. Certified Diabetes Educator

- a. On the Provider Login Screen, log in using the username and password provided by the research team on the Patients Screen.
- b. Choose patient Will Owens on the Visit Status Screen.
- c. Add comments needs to be followed up regarding ketosis education in the comments for provider text box on the Visit Status Screen.
- d. Add a goal for the patient log out of Goals-to-Guide application.

After the tasks were performed, an informal semi-structured interview was conducted with each participant to explore their experience with the GTG application. The interview looked at how the participants thought the application could be improved and what their thoughts were about the overall

benefit of such an application. The interview asked the following questions, all of which were elaborated on.

- 1. How long have you been a patient of this clinic?
- 2. What were some of the strengths of the GTG app? Why?
- 3. What were some of the weaknesses of the GTG app? Why?
- 4. What was the hardest task to perform on the app?
- 5. Have you used apps to manage T2D before?
- 6. Do you have any concerns regarding the app?

Finally, the participants were asked to complete a questionnaire to further elaborate on their experience with the GTG application. The questionnaire asked the participants to rate their experience with the GTG application on a scale from 1 to 6 (1= I strongly disagree, 6= I completely agree) against the following criterion:

- 1. Guide to Goals will motivate users to increase frequency of incorporating best practices for managing Type 2 Diabetes.
- 2. Guide to Goals is a user friendly application.
- 3. Guide to Goals will facilitate conversation between the various members of the care team.
- 4. Guide to Goals was easy to use for the first time.
- 5. I will feel comfortable using Guide to Goals during a real visit at Children's Healthcare of Atlanta